CLINICAL TRIAL: NCT04727073
Title: Spironolactone in the Treatment of Heart Failure- a Double-blind, Randomized, Placebo-controlled, Parallel Group Interventional Phase III Study to Determine Efficacy and Safety of Spironolactone on the Composite Endpoint of Recurrent Heart Failure Hospitalizations and Cardiovascular Death in Patients with Heart Failure with Mid-range or Preserved Ejection Fraction
Brief Title: Spironolactone in the Treatment of Heart Failure
Acronym: SPIRIT-HF
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: No extension of study funding by the DZHK following COVID-19 pandemic-induced prolongation of the recruitment period, also requiring manufacturing of further study drug batches
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Deutsches Zentrum für Herz-Kreislauf-Forschung (DZHK) (Other); Echo Core Lab Berlin (Unknown); University of Göttingen (Other); University Medicine Greifswald (Other); Ludwig-Maximilians - University of Munich (Other); Institute for Cardiovascular Computer-assisted Medicine, Charité (Unknown); Coordinating Centre for Clinical Trials, Charité (Unknown)
Responsible Party: Principal Investigator, Univ.-Prof. Dr. med. Frank Edelmann, Univ. Prof. Dr. med. Frank Edelmann, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SPIRIT-HF DZHK08; SPIRIT-HF DZHK8 (Other Grant/Funding Number: Deutsches Zentrum für Herzkreislaufforschung)
Record Dates: First submitted 2019-01-28; First posted 2021-01-27 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Heart Failure with Mid-range Ejection Fraction; Heart Failure with Preserved Ejection Fraction
Keywords: heart failure; mid-range ejection fraction; preserved ejection fraction; diastolic dysfunction; Spironolactone; Mineralcorticoid Receptor Antagonist
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (Experimental): Experimental: Spironolactone Spironolactone (an aldosterone antagonist) in tablet form taken daily. The initial study drug dose is 25 mg/day (one tablet) and may be titrated up to 50 mg/day (two tablets) within 4 weeks if kidney function at VR was > 30 mL/min/m2 and potassium < 4.5 mmol/L.
  Interventions: Drug: Experimental: Spironolactone
- Arm B (Placebo Comparator): Placebo Comparator: Placebo Placebo of Spironolactone in tablet form taken daily with dosage escalation rules in accordance with dosage of the study drug Spironolactone.
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: Experimental: Spironolactone — Spironolactone (an aldosterone antagonist) in tablet form taken daily. The initial study drug dose is 25 mg/day (one tablet) and may be titrated up to 50 mg/day (two tablets) within 4 weeks if kidney function at VR was > 30 mL/min/m2 and potassium < 4.5 mmol/L.
  Arms: Arm A
Drug: Placebo Comparator — Placebo of Spironolactone in tablet form taken daily with dosage escalation rules in accordance with dosage of the study drug Spironolactone.
  Arms: Arm B

SUMMARY:
The purpose of this study is to determine whether the treatment of patients with HFmrEF and HFpEF at high risk of cardiovascular events with the mineralocorticoid receptor antagonist (MRA) spironolactone reduces a composite of recurrent heart failure hospitalizations and cardiovascular mortality.

DETAILED DESCRIPTION:
The primary objective of the SPIRIT-HF study is to compare Spironolactone to Placebo in reducing the rate of the composite endpoint of recurrent heart failure hospitalizations and cardiovascular (CV) death in symptomatic HF patients (NYHA II-IV) with mid-range (LVEF 40- 49 %) or preserved (LVEF ≥ 50 %) ejection fraction.

The efficacy and safety of mineralocorticoid receptor antagonist (MRA) in reducing the risk of death and hospitalizations has been proven with two separate substances (Spironolactone; RALES 1999 and Eplerenone; EMPHASIS 2011) in symptomatic heart failure patients with reduced left- ventricular ejection fraction (HFrEF). In 2013 the TOPCAT investigators tried to proof similar efficacy in patients with heart failure and preserved ejection fraction (≥ 45%). Because of regional variations in the enrollment process and difficulties regarding drug adherence the trial revealed neutral findings but the substance spironolactone was still able to show its potential benefit in the American cohort. Hence, the investigators see a strong rationale for testing a mineralocorticoid receptor blocker in patients suffering from heart failure with mid-range or preserved left ventricular ejection fraction.

Intervention:

Mineralocorticoid receptor blocker Spironolactone in tablet form taken daily. Starting dosage will be 25 mg OD with dosage escalation to 50 mg OD within 4 weeks if kidney function at VR was > 30 mL/min/m2 and potassium < 4.5 mmol/L. Spironolactone is not approved for the treatment of HFmrEF and HFpEF.

Matching placebo in tablet form taken daily with dosage escalation rules in accordance with dosage of the study drug Spironolactone.

Visits:

Screening (VScr), Visit of Randomization (VR), V1 Safety Visit (1 week), V2 (4 weeks), V2S Safety Visit (5 week), V3 (4 months), V4 (8 months), V5 (12 months), V6 (18 months), V7 (24 months), V8 (30 months), V9 (36 months), V10 (42 months), V11/EOT (48 months); VXS (1 week after Visit X).

Individual intervention duration with spironolactone or placebo will be continued until the overall expected event rate is reached or until withdrawal of informed consent. Based on previous HF trials the investigators calculate a mean follow-up duration of 3 years (range 2-4 years) depending on the individual inclusion date.

Duration of follow-up will be event-rate based, with an expected overall study duration of 60 months. With an anticipated recruitment phase of 24 months; this will result in a maximum follow-up of 48 months and an average follow-up per patient of 36 months assuming a constant recruitment rate.

ELIGIBILITY:
Inclusion Criteria:

Patients eligible for inclusion in this study have to fulfill all of the following criteria:

1. Written informed consent.
2. Male or female, age ≥ 50 years
3. Current symptoms of Heart Failure (NYHA ≥ II) during VR
4. Symptom(s) of HF ≥ 30 days prior to VR
5. HF Hospitalization or treatment with intravenous (IV) diuretics for worsening HF within 12 months prior to VR
6. Left ventricular ejection fraction ≥ 40 % at screening measured by echocardiography and evidence of structural/ functional abnormalities (at least one of the following criteria): LAVI > 34 ml/m2// E/émean ≥ 13// Mean e' (septal and lateral) < 9 cm/s
7. NT-proBNP > 300 pg/ml (SR) or > 900 pg/ml (AF) on the Visit 1 ECG; only if NT-proBNP is NOT available: BNP > 80/ 250 pg/ml (SR/AF)
8. Controlled systolic BP: defined as a target systolic BP < 140 mm Hg. Subjects with BP up to and including 160 mm Hg are eligible for enrollment if on 3 or more medications to control BP (Patients with uncontrolled BP should be considered for Re-Screening after optimization of antihypertensive therapy has been established)
9. Serum potassium < 5.0 mmol/L prior to randomization

Exclusion Criteria:

Patients fulfilling any of the following criteria are not eligible for inclusion in this study. The investigator may apply no additional exclusion criteria, in order to ensure that the study population will be representative of all eligible patients.

1. Hyperkalemia (potassium level ≥ 5.5 mmol/L) within the past two weeks before VR
2. Hyponatraemia (sodium level < 135 mmol/L) prior to randomization
3. Severe renal dysfunction, defined as an estimated glomerular filtration rate of less than 30 mL/min/1.73m2) as calculated by the Modification in Diet in Renal Disease (MDRD) formula at Visit 1 or serum creatinine level ≥ 1,8 mg/dl (> 160 μmol/ml)
4. History of anuria or acute renal failure (as defined by the RIFLE criteria for AKI; see Appendix XVIII.3) within the past two weeks before VRenal dysfunction, defined as an estimated glomerular filtration rate of less than 30 mL/min/1.73m2) as calculated by the Modification in Diet in Renal Disease (MDRD) formula at VScr/VR or serum creatinine level ≥ 1,8 mg/dl (> 160 μmol/ml)History of anuria or acute renal failure (as defined by the RIFLE criteria for AKI; see Appendix XVIII.3) within the past two weeks prior to randomization
5. Acute coronary syndrome (including MI) and elective PCI within 30 days prior to VR.
6. Cardiac surgery, other major CV surgery, or urgent percutaneous coronary intervention (PCI) within the 3 months prior to VR
7. Current acute decompensated HF requiring augmented therapy with i.v. diuretics, i.v. vasodilators and/or i.v. inotropic drugs. Patients are eligible after initial stabilization.
8. Probable alternative diagnoses that in the opinion of the investigator could account for the patient's HF symptoms (i.e., dyspnea, fatigue) such as significant pulmonary disease (including primary pulmonary HTN), anemia or obesity. Specifically, patients with the following are not eligible for randomization:

   * Severe pulmonary disease including chronic obstructive pulmonary disease (COPD) or severe asthma bronchiale ( (ie requiring home oxygen, chronic nebulizer therapy, chronic oral steroid therapy) or
   * anemia (hemoglobin < 10 g/dL males and < 9.5 g/dL females), or
   * body mass index (BMI) > 40 kg/m2
9. Evidence of right sided HF in the absence of left-sided structural heart disease.
10. Specific etiologies such as infiltrative, genetic hypertrophic cardiomyopathy, pericardial constriction, sarcoidosis, amyloidosis and any other storage diseases.
11. Clinically significant congenital heart disease underlying heart failure.
12. Life-threatening or uncontrolled dysrhythmia, including symptomatic or sustained ventricular tachycardia and uncontrolled persistent or permanent atrial fibrillation (AF) or flutter (with a heart rate > 100 beats per minute (bpm), RACE II) during VR. If AF with HR > 100/min, the patient may be rescreened after treatment for rate control.
13. Presence of significant (i.e., more than moderate) valvular heart disease expected to lead to surgery during the trial in the investigators opinion.
14. Stroke, transient ischemic attack, carotid surgery or carotid angioplasty within the 3 months prior to VR.
15. Coronary or carotid artery disease or valvular heart disease likely to require surgical or percutaneous intervention within the 6 months after VR in the investigators opinion.
16. Patients with prior major organ transplant or intent to transplant (on transplant list) or with current ventricular assist device (VAD) therapy.
17. Evidence of hepatic disease as determined by any one of the following: SGOT (AST) or SGPT (ALT) values exceeding 3x the upper limit of normal (ULN), bilirubin >1.5 mg/dl at VR.
18. Evidence of present bilateral renal artery stenosis
19. Known intolerance or history of hypersensitivity to the active substance (Spironolactone) or to any of the excipients of the Investigational Medicinal Product (IMP) or placebo.
20. Present use of any aldosterone antagonist, potassium supplements or potassium sparing diuretics at the time of enrollment. (Consider stopping these potassium sparing drugs if clinically possible and upon discussion with the patient)
21. Required treatment with prohibited Co-medications according to the summary of product characteristics with the exception of ACE inhibitors or angiotensin receptor blockers (as described in the protocol in IV.2).

    , careful monitoring of plasma lithium and dose adjustment are required.
22. Use of other investigational drugs at the time of enrollment, or within 30 days or 5 half-lives before enrollment, whichever is longer.
23. Any condition that, in the opinion of the investigator may prevent the subject from adhering to the study protocol (e.g. history of non-compliance to medical regimens, patients who are considered potentially unreliable, patients with a history of addiction).
24. History or presence of any other disease (i.e. including malignancies) with a life expectancy of < 1 years.
25. History of non-compliance to medical regimens and patients who are considered potentially unreliable.
26. Subjects who are legally detained in an official institution.
27. Subjects who may be dependent on the sponsor, the investigator or the trial sites, have to be excluded from the trial.
28. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin (hCG) laboratory test.
29. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during study participation and until 2 months after the last dose off study drug.

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 743 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Primary Objective: Cumulative number of primary composite events of cardiovascular (CV) death and total HF hospitalizations | Time Frame: Total follow up time (up to 48 months)
  Cumulative number of primary composite events of cardiovascular (CV) death and total (first and recurrent) HF hospitalizations in symptomatic HF patients (NYHA II-IV) with mid-range (LVEF 40- 49 %) or preserved (LVEF ≥ 50 %) ejection fraction.

SECONDARY OUTCOMES:
Secondary Objective: Comparison of spironolactone to placebo in reducing the rate of hospitalisations and deaths | Time Frame: Total follow up time (up to 48 months)
  * To compare Spironolactone to placebo in reducing the recurrent rate of heart failure Hospitalizations [Time Frame: Follow-up time up to 48month.]
  * To compare Spironolactone to placebo in reducing the rate of recurrent non-fatal hospitalizations from cardiovascular (CV) cause (i.e. hospitalization for non-fatal MI, non-fatal stroke, or the management of heart failure, whichever occurred first) [Time Frame: Total follow up time (up to 48 months)].
  * To compare Spironolactone to placebo in reducing the recurrent rate of hospitalizations from any cause [Time Frame: Total follow up time (up to 48 months)].
  * To compare Spironolactone to placebo in reducing the rate of death from cardiovascular (CV) cause [Time Frame: Total follow up time (up to 48 months)].
  * To compare Spironolactone to placebo in reducing the rate of death from any cause [Time Frame: Total follow up time (up to 48 months)].

CONTACTS AND LOCATIONS:
Overall Officials: Burkert Pieske, Prof. MD, Principal Investigator — Charité University of Medicine
Locations (69):
- Austria (5):
  - Medical University of Graz, Graz
  - Medical University Innsbruck, Innsbruck
  - Clinic Klagenfurt Wörthersee, Klagenfurt
  - University Hospital St. Pölten, Pölten
  - Medical University of Vienna, Vienna
- France (10):
  - Besançon University Hospital, Besançon
  - Centre Hospitalier de Beziers, Béziers
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - Groupe Hospitalier de la Rochelle-Ré-Aunis, La Rochelle
  - CHU Grenoble Alpes Hopital Michallon, La Tronche
  - CHU Arnaud de villeneuve, Montpellier
  - CHRU Nancy Brabois, Nancy
  - CHU Haut Lévêque Cardiologie, Pessac
  - Hôpital Sainte Musse, Toulon
  - CHU Toulouse - Hôpital Rangueil, Toulouse
- Germany (38):
  - Kardiologische Praxis Dr. Wolfgang Jungmair, Bad Homburg
  - Kerckhoff Heart and Thorax Center, Bad Nauheim
  - Herz- und Diabeteszentrum NRW, Bad Oeynhausen, Bad Oeynhausen
  - Charité University of Medicine Berlin, CCM, Berlin
  - Klinische Forschung Berlin GbR, Berlin
  - Studienzentrum Rankestraße, Berlin
  - Charité University of Medicine, CBF, Berlin
  - Caritas-Klinik Maria Heimsuchung, Berlin
  - Charité University of Medicine (CVK), Berlin
  - German Heart Center Berlin, Clinic for Internal Medicine - Cardiology, Berlin
  - Helios Klinikum Emil von Behring GmBH, Berlin
  - Städtisches Klinikum Brandenburg GmbH, Brandenburg
  - Stiftung Bremer Herzen (BIHKF), Bremen
  - Zentrum für klinische Studien Dresden, Dresden
  - Heart Center Dresden, Technical University of Dresden, Dresden
  - Zentrum für klinische Studien Südbrandenburg, Elsterwerda
  - University Hospital of Giessen, Giessen
  - University of Goettingen, Goettigen
  - University Medicine Greifswald, Greifswald
  - Universitätsklinikum Halle (Saale), Halle
  - University Heart Center Hamburg, Hamburg
  - University of Heidelberg, Heidelberg
  - University Hospital Jena, Jena
  - University Medical Center of Schleswig-Holstein, Campus Kiel, Kiel
  - Universitätsklinikum Leipzig, Leipzig
  - Heart Center Leipzig-University Hospital, Leipzig
  - University Hospital Schleswig-Holstein, University Heart Centre Lübeck, Lübeck
  - University Hospital Mainz, Mainz
  - University Medical Center Mannheim, Medical Faculty Mannheim, Heidelberg University, Mannheim
  - Kliniken Maria Hilf GmbH, Mönchengladbach
  - German Heart Center Munich, Munich
  - University Hospital Klinikum rechts der Isar (TUM), Munich
  - University Hospital Munich, Ludwig-Maximilians University, Munich
  - University Hospital rechts der Isar, Munich
  - Kardiologische Praxis Am Park Sanssoucci, Potsdam
  - Praxis Dr. Markus Knapp/Daniela Breuninger, Schwäbisch Hall
  - MVZ Schwering West GmbH, Schwerin
  - Universitätsklinikum Ulm, Ulm
- Netherlands (7):
  - Meander Medisch Centrum, Amersfoort
  - Ziekenhuis Amstelland, Amstelveen
  - OLVG locatie Oost, Amsterdam
  - Van Weel-Bethesda Ziekenhuis, Dirksland
  - St. Jansdal Ziekenhuis, Harderwijk
  - Elkerliek Ziekenhuis, Helmond
  - Gelre Ziekenhuizen, Zutphen
- Serbia (9):
  - Institute for Rehabilitation, Belgrade
  - Clinical Hospital Center B. Kosa, Belgrade
  - Clinical Hospital Center Dr. Dragisa Misovic, Belgrade
  - Clinical Hospital Center Zvezdara, Belgrade
  - Dedinje Cardiovascular Institute, Belgrade
  - Insitute of Cardiovascular Diseases of Vojvodina, Kamenitz
  - Nis Clinical Center, Niš
  - General Hospital Uzice, Užice
  - General Hospital Vršac, Vršac

IPD SHARING:
Plan to Share IPD: No